CLINICAL TRIAL: NCT01271894
Title: The Intensive Pharmacokinetics Sub-study of Encore1: A Randomised, Double-blind, Placebo-controlled, Clinical Trial to Compare the Safety and Efficacy of Reduced Dose Efavirenz (EFV) With Standard Dose EFV Plus Two Nucleotide Reverse Transcriptase Inhibitors (N(t)RTI) in Antiretroviral-naïve HIV-infected Individuals Over 96 Weeks
Brief Title: The Intensive Pharmacokinetics Sub-study of Encore1 (ENCORE1-PK)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: NCHECR-ENCORE1-PK
Record Dates: First submitted 2011-01-05; First posted 2011-01-07 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2012-11

CONDITIONS: HIV Infection
Keywords: HIV; efavirenz; pharmacokinetic
MeSH Terms: conditions — HIV Infections | interventions — efavirenz

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reduced dose Efavirenz arm (Experimental): Participants randomized in main study to receive EFV (400 mg once daily; 2 x 200 mg + 1 x placebo once daily) plus tenofovir/emtricitabine (300/200 mg) fixed-dose combination once daily
  Interventions: Drug: Efavirenz
- Normal Efavirenz dose arm (Active Comparator): Patients randomized in the main study to receive EFV (600 mg once daily; 3 x 200 mg once daily) plus tenofovir/emtricitabine (300/200 mg) fixed-dose combination once daily
  Interventions: Drug: Efavirenz

INTERVENTIONS:
Drug: Efavirenz — 600 mg once daily; given as 3 x 200 mg once
  Arms: Normal Efavirenz dose arm
Drug: Efavirenz — 400 mg once daily; given as 2 x 200 mg + 1 x placebo
  Arms: Reduced dose Efavirenz arm

SUMMARY:
Safety and efficacy are key issues in antiretroviral therapy (ART) selection. Efavirenz (EFV) is an important component of combination ART in treatment naive individuals. Like many drugs, there are inter-individual differences in the efficacy and tolerability of EFV. The Encore1 study provides an opportunity to examine the pharmacokinetics (PK)(processes by which a drug is absorbed, distributed, metabolized, and eliminated by the body) of EFV in blood samples collected over a 24-hour dosing interval in participants receiving either standard 600 mg or reduced 400 mg dose EFV once daily.

DETAILED DESCRIPTION:
This sub-study will investigate the relationships between dosage, EFV plasma concentrations, toxicity and virological efficacy. EFV concentrations in dried blood spots and matched plasma and will be evaluated to determine the utility of dried blood spot measurements in measuring EFV plasma concentrations. Measurements dried blood spots could potentially be a cheap and easy alternative to measurements in plasma. Dried blood spots can be easily collected from venous blood or fingerprick, do not need plasma separation and potentially need less stringent storage conditions during shipment.

ELIGIBILITY:
All participants enrolled into the main Encore1 study at participating sub-study sites will be eligible to participate.

Participants must meet the following additional inclusion criteria prior to intensive pharmacokinetic assessment. Inclusion Criteria:

* provide written sub-study consent at or before week 0
* taken randomized study drugs for at least 4 weeks but less than 8 weeks
* taken EFV in the evening for at least 7 days
* taken all EFV doses over the 3 preceding days.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
To compare the pharmacokinetic parameters of EFV determined from blood collected over a 24-hour dosing interval in blinded samples from participants taking either 600 mg or 400 mg once daily in combination with Truvada. | 48 weeks

SECONDARY OUTCOMES:
To compare the safety and tolerability of EFV 400 mg versus 600 mg given once daily. | 48 weeks
To investigate the correlation between EFV concentration measurements from dried blood spots and concentration measured in matched plasma samples. | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, Dr., Principal Investigator — Chelsea & Westminster Hospital
Locations (4):
- Hospital J.M. Ramos Mejia, Buenos Aires, Argentina
- Desmond Tutu HIV Foundation, Cape Town, South Africa
- Thai Red Cross-AIDS Research Centre, HIV-NAT Research Collaboration, Bangkok, Thailand
- Chelsea and Westminister Hospital, London, United Kingdom